CLINICAL TRIAL: NCT01553526
Title: BIOTRONIK - Safety and Performance Registry for an All-comers Patient Population With the Limus Eluting Orsiro Stent System Within Daily Clinical Practice - III
Brief Title: BIOFLOW-III All-comers Orsiro Safety and Performance Registry
Acronym: BIOFLOW-III
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: C1101
Record Dates: First submitted 2012-03-08; First posted 2012-03-14 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia
Keywords: International; Multicenter; Observational registry; All-comers open label registry; Orsiro Drug Eluting Stent (DES); Stenting; Treatment of Coronary Artery Disease; Coronary revascularization; Percutaneous Coronary Intervention; STEMI; NSTEMI; Ischemia; Angina; Subgroups; Acute Myocardial Infarction; Diabetes; Small Vessels; Chronic Total Occlusion (CTO)
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Ischemia; Angina Pectoris; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Orsiro DES

SUMMARY:
This registry is a clinical post-market evaluation of the Orsiro LESS in subjects requiring coronary revascularization with Drug Eluting Stents (DES).

DETAILED DESCRIPTION:
For the majority of Coronary Artery Disease (CAD), treatment with Percutaneous Transluminal Coronary Angioplasty (PTCA) provides high initial procedural success. However, the medium to long-term complications range from rather immediate elastic recoil or vessel contraction to longer processes like smooth muscle cell proliferation and excessive production of extra cellular matrix, thrombus formation and atherosclerotic changes like restenosis or angiographic re-narrowing. The reported incidence of restenosis after PTCA ranges from 30%-50%. Such rates of recurrence have serious economic consequences.

Bare Metal Stents (BMS), designed to address the limitations of PTCA, reduced the angiographic and clinical restenosis rates in de novo lesions compared to PTCA alone and decreased the need for CABG. BMS substantially reduced the incidence of abrupt artery closure, but restenosis still occurred in about 20%-40% of cases, necessitating repeat procedures.

The invention of Drug Eluting Stents (DES) significantly improved on the principle of BMS by adding an antiproliferative drug (directly immobilised on the stent surface or released from a polymer matrix), which inhibits neointimal hyperplasia. The introduction of DES greatly reduced the incidence of restenosis and resulted in a better safety profile as compared to BMS with systemic drug administration.

These advantages and a lower cost compared to surgical interventions has made DES an attractive option to treat coronary artery disease. This observational registry is designed to investigate and collect clinical evidence for the clinical performance and safety of the Orsiro Drug Eluting Stent System in an all-comers patient population in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic coronary artery disease
* Subject has signed informed consent for data release
* Subject is geographically stable and willing to participate at all follow-up assessments
* Subject is ≥ 18 years

Exclusion Criteria:

* Subject did not sign informed consent for data release
* Pregnancy
* Known intolerance to aspirin, clopidogrel, ticlopidine, heparin or any other anticoagulation / antiplatelet therapy required for PCI, stainless steel, Sirolimus or contrast media
* Planned surgery within 6 months of PCI unless dual antiplatelet therapy will be maintained
* Currently participating in another study and primary endpoint is not reached yet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers patient population with all subjects requiring coronary revascularization with a Drug Eluting Stent (DES)
Sampling Method: Non-Probability Sample
Enrollment: 1356 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  Composite of cardiac death, target vessel Q-wave or non-Q wave Myocardial Infarction (MI), Emergent Coronary Artery Bypass Graft (CABG), clinically driven Target Lesion Revascularization (TLR)

SECONDARY OUTCOMES:
Target Lesion Failure (TLF) | 6, 36 and 60 months
Target Vessel Revascularization (TVR) | 6, 12, 36 and 60 months
  Any repeat revascularization of the target vessel.
Target Lesion Revascularization (TLR) | 6, 12, 36 and 60 months
  Any repeat revascularization of the target lesion.
Stent Thrombosis | 6, 12, 36 and 60 months
Clinical Device Success | At time of intervention
Clinical Procedural Success | During the hospital stay to a maximum of the first seven days post index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Esther Gerteis, Study Director — Biotronik AG; Johannes Waltenberger, Prof., Principal Investigator — University Hospital Muenster
Locations (43):
- University Hospital Innsbruck, Innsbruck, Austria
- Clinica Tabancura, Santiago, Chile
- Gentofte Universitets Hospital, Hellerup, Denmark
- France (9):
  - Clinique Rhone Durance, Avignon
  - CHU Bocage Dijon, Dijon
  - CCML Le Plessis Robinson, Le Plessis-Robinson
  - CHRU Brabois Nancy, Nancy
  - CH Niort, Niort
  - Clinique Saint Hilaire Rouen, Rouen
  - CHRU Rangueil Toulouse, Toulouse
  - CHG Troyes, Troyes
  - CH Valence, Valence
- Germany (14):
  - Segeberger Kliniken, Bad Segeberg
  - Klinikum im Friedrichshain, Berlin
  - Kardiologisch-Angiologische Praxis Hegeler, Bremen
  - Klinikum Coburg, Coburg
  - Krankenhaus Martha Maria gGmbH, Klinik fuer Innere Medizin I, Halle
  - Asklepiosklinik St. Georg, Hamburg
  - Uniklinik Heidelberg, Medizinische Uniklinik, Heidelberg
  - Klinikum Landshut-Achdorf Medizinische Klinik I, Landshut
  - University of Leipzig, Leipzig
  - LMU-Großhadern, Munich
  - HZ Muenchen-Bogenhausen, Klinik fuer Kardiologie und Internistische Intensivmedizin, Munich
  - Universitaetsklinikum Muenster, Münster
  - Uniklink Regensburg, Regensburg
  - Kliniken Villingen - Kardiologie, Villingen-Schwenningen
- Italy (2):
  - Centro cardiologico Monzino, Milan
  - Cattedra Universitaria, Divisione Cardiologia, Policlinico Tor Vergata, Rome
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga Eastern Clinical University Hospital, Riga
- Netherlands (6):
  - VU Medical Center HV Amsterdam, Amsterdam
  - Alysis Hospital, Arnhem
  - Amphia Ziekenhuis Breda, Breda
  - St. Antonius Ziekenhuis, Nieuwegein
  - ZorgSaam Terneuzen, Terneuzen
  - Twee Steden Hospital Tilburg, Tilburg
- Centro Hospitalar de Coimbra, São Martinho do Bispo, Portugal
- Hospital de Navarra, Pamplona, Spain
- Universitetssjukhuset Oerebro, Kardiologiska Kliniken, Örebro, Sweden
- Switzerland (2):
  - Clinique Cecil, Lausanne
  - Kantonsspital Liestal, Liestal
- United Kingdom (2):
  - Craigavon Area Hospital Lurgan Road Co. Armagh, Northern Ireland, Belfast
  - The Heart Hospital, UCLH, London

REFERENCES:
- [Derived] Toelg R, Slagboom T, Waltenberger J, Lefevre T, Saito S, Kandzari DE, Koolen J, Richardt G. Individual patient data analysis of the BIOFLOW study program comparing safety and efficacy of a bioresorbable polymer sirolimus eluting stent to a durable polymer everolimus eluting stent. Catheter Cardiovasc Interv. 2021 Nov 1;98(5):848-856. doi: 10.1002/ccd.29254. Epub 2020 Sep 5. PMID 32890442
- [Derived] Waltenberger J, Brachmann J, van der Heyden J, Richardt G, Frobert O, Seige M, Friedrich G, Erglis A, Winkens M, Hegeler-Molkewehrum C, Neef M, Hoffmann S; BIOFLOW-III Investigators. Five-Year Results of the Bioflow-III Registry: Real-World Experience with a Biodegradable Polymer Sirolimus-Eluting Stent. Cardiovasc Revasc Med. 2020 Jan;21(1):63-69. doi: 10.1016/j.carrev.2019.03.004. Epub 2019 Mar 15. PMID 30922870
- [Derived] Waltenberger J, Brachmann J, van der Heyden J, Richardt G, Frobert O, Seige M, Erglis A, Dewilde W, Winkens M, Hegeler-Molkewehrum C, Klein N, Hoffmann S; BIOFLOW-III Investigators. Real-world experience with a novel biodegradable polymer sirolimus-eluting stent: twelve-month results of the BIOFLOW-III registry. EuroIntervention. 2016 Feb;11(10):1106-10. doi: 10.4244/EIJY15M03_08. PMID 25782184